CLINICAL TRIAL: NCT05769829
Title: ImmuneSense™ IBD Study
Status: Terminated | Type: Observational
Why Stopped: Enrollment challenges for cohort 2
Sponsor: Adaptive Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-01038
Record Dates: First submitted 2023-01-11; First posted 2023-03-15 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; Ulcerative colitis; Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Pre-diagnosis/+Gastrointestinal Symptoms: Up to 450 participants with gastrointestinal symptoms, undergoing endoscopy with biopsy will have blood drawn, metadata collected, and tissue from endoscopy collected for analysis. Additional blood draws at various timepoints during the study; at follow up visits, at time of flare, medication change, surgery, or repeat endoscopy.
  In addition to the 450 participants enrolled, 50 more participants that meet inclusion/exclusion for cohort 1 will be enrolled to complete only the initial visit and endoscopy visit. Participants will have blood drawn, metadata collected, and tissue from endoscopy collected for analysis.
- Cohort 2: Diagnosed Inflammatory Bowel Disease, Pre-treatment: Up to 400 participants recently diagnosed with inflammatory bowel disease but not yet started on a medication regimen to address their symptoms will have blood drawn with metadata attached. Additional blood draws at various timepoints during the study; at follow up visits, at time of flare, medication change, surgery, or repeat endoscopy.
- Cohort 3: Potential Cross-Reactive Diseases: Patients will be eligible for this cohort if they fail to be diagnosed with inflammatory bowel disease but have a confirmed diagnosis of potential cross reactive disease states including Irritable Bowel Syndrome, Functional Diarrhea, Celiac Disease.
- Cohort 4: Healthy Controls: Up to 228 participants free from GI symptoms for the last 90 days and no previous medical history or clinical diagnosis of GI illness.

SUMMARY:
This study will enroll adult and pediatric participants across 3 phases: Research phase, Clinical Validation (CV) and Analytical Validation (AV) phase.

Sites selected to participate in the study will enroll participants in the either the Research phase or CV and AV phase. Research Phase will enroll participants in Cohort 1 Pre-diagnosis/+GI symptoms only.

CV and AV phase will be open to enrollment in parallel. CV phase will enroll participants in Cohort 2 Diagnosed IBD, Pre-treatment, Cohort 3 Potential Cross-Reactive Diseases and Cohort 4 Healthy controls.

AV phase will enroll participants in Cohort 2 Diagnosed IBD, Pre-treatment and Cohort 4 Healthy controls. Enrollment will be ongoing until sponsor notification for closure.

ELIGIBILITY:
Cohort 1: Pre-diagnosis/+GI symptoms Inclusion criteria

* i.GI symptoms with clinical suspicion for inflammation and planned for endoscopy at discretion of clinician
* ii. Male and female participants of any race and ethnicity between 7 to 89 years of age (inclusive) at the time of enrolling in the study
* iii. Must be able to communicate with the investigator, understand and comply with the requirements of the study

Exclusion Criteria

* Age <7 years or >89 years
* Known IBD (Ulcerative colitis, Crohn's disease, indeterminate colitis) and Celiac
* Known active malignancy
* Active Hepatitis B, C or HIV infection(s)
* Use of systemic high dose corticosteroids (above 20mg/day prednisone by mouth) within 30 days prior to the blood draw
* Protected populations including pregnant women, prisoners, mentally disabled persons, and wards-of-the state
* Any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study
* Donated more than 500cc or 1 pint of blood in the past 60 days prior to the blood draw (at the discretion of the investigator)

Cohort 2: Diagnosed IBD, Pre-treatment Inclusion criteria

* Diagnosis of Crohn's disease or Ulcerative colitis made with endoscopy (within 6 months), clinical, imaging, and histological findings.
* Male and female participants of any race and ethnicity between 7 to 89 years of age (inclusive) at the time of enrolling in the study
* Must be able to communicate with the investigator, understand and comply with the requirements of the study

Exclusion Criteria

* Age <7 years or >89 years
* Known active malignancy
* Known Celiac disease
* Active Hepatitis B, C or HIV infection(s)
* Active gastrointestinal infection within 30 days prior to enrollment
* Protected populations including pregnant women, prisoners, mentally disabled persons, and wards-of-the state
* Any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study
* Donated more than 500cc or 1 pint of blood in the past 60 days prior to the blood draw (at the discretion of the investigator)
* On any treatment for IBD- systemic corticosteroids within 30 days, immunomodulator, 5-ASA, biologic therapy
* Plan to initiate therapy as part of a clinical trial of a non-FDA-approved IBD therapy

Cohort 3: Potential Cross-Reactive Disease States Inclusion criteria

* Confirmed, documented diagnoses for one of the following diseases:
* Irritable Bowel Syndrome, Functional Diarrhea (Endoscopy negative for inflammation)
* Celiac disease (Serology positive (ttg IgA+) AND Upper endoscopy confirming Celiac disease diagnosis)
* Diverticulitis, and other forms of microscopic colitis
* Infectious etiologies: E. coli, Klebsiella pneumoniae, Salmonella spp., Shigella spp., Yersinia spp (Positive stool culture or PCR)
* For infections, active infections are required or within 30 days of infection.
* Male and female participants of any race and ethnicity between 7 to 89 years of age (inclusive) at the time of enrolling in the study
* Must be able to communicate with the investigator, understand and comply with the requirements of the study

Exclusion Criteria

* Age <7 years or >89
* Individuals with a prior or current clinical diagnosis of IBD
* Active Hepatitis B, C or HIV infection(s)
* Protected populations including pregnant women, prisoners, mentally disabled persons, and wards-of-the state
* Any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study
* Donated more than 500cc or 1 pint of blood in the past 60 days prior to the blood draw (at the discretion of the investigator)

Cohort 4: Healthy Controls Inclusion criteria

* Male and female participants of any race and ethnicity between 7 to 89 years of age (inclusive) at the time of enrolling in the study
* Must be able to communicate with the investigator, understand and comply with the requirements of the study Exclusion criteria
* Age <7 years or >89
* GI symptoms in last 90 days (Abdominal pain, diarrhea, blood in stool, weight loss, vomiting)
* Individuals with a prior or current clinical diagnosis of IBD, Celiac disease, active infection
* Family history of Crohn's disease, indeterminate colitis or ulcerative colitis
* Active Hepatitis B, C or HIV infection(s)
* Protected populations including pregnant women, prisoners, mentally disabled persons, and wards-of-the state
* Any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study
* Donated more than 500cc or 1 pint of blood in the past 60 days prior to the blood draw (at the discretion of the investigator)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Pre-diagnosis/+Gastrointestinal Symptoms Participants with gastrointestinal symptoms, undergoing endoscopy with biopsy will have blood drawn, metadata collected, and tissue from endoscopy collected for analysis.
  Cohort 2: Diagnosed Inflammatory Bowel Disease, Pre-treatment Participants recently diagnosed with IBD but not yet started on a medication regimen to address their symptoms will have blood drawn with metadata attached.
  Cohort 3: Potential Cross-Reactive Diseases Participants with confirmed diagnosis of potential cross reactive disease states including Irritable Bowel Syndrome, Functional Diarrhea, Celiac Disease.
  Cohort 4: Healthy Controls Participants free from GI symptoms for the last 90 days and no previous medical history or clinical diagnosis of GI illness.
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of T-Detect IBD | Initial Study visit/Baseline
  To evaluate the sensitivity and specificity of T-Detect IBD, by interrogating the peripheral T cell repertoire for TCRs enhanced in IBD, to aid in diagnosis of IBD.
  To evaluate the sensitivity and specificity of T-Detect IBD relative to endoscopy with biopsies.
  To evaluate the sensitivity and specificity of T-Detect IBD as a prognostic marker for medication response.

SECONDARY OUTCOMES:
Future/Additional research | Initial Study visit/Baseline
  Samples not allocated to primary objective may be used for additional research and/or development, and clinical and analytical development/validation efforts may utilize samples collected from this study.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Hope Clinic & Research Center LLC, Hialeah, Florida
  - Gold Coast Health Research Center, LLC, Miami, Florida
  - Sanitas Research, Miami, Florida
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastroenterology Consultants of South Texas, PA, Brownsville, Texas